CLINICAL TRIAL: NCT04081870
Title: IS Three d Power Doppler of the Endometrial and Subendometrial Regions Effective?
Brief Title: IS Three d Power Doppler of the Endometrial and Subendometrial Regions Effective in Predicting Endometrial Implantation?
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, khalid mohammed salama, principal investigator, Benha University
Other Study IDs: khalid 6
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Infertility
Keywords: doppler,endometrial,implantation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICSI cases: All women underwent long agonist protocol for controlled ovarian hyperstimulation The GnRH agonist was started in the previous mid-luteal phase . After the confirmation of pituitary down regulation , the HMG ampoules were started by 225 IU/day . During the follow up of overstimulation, the doses were adjusted according to the response of patient. All women underwent serial TVS until at least three dominant follicles were reached in every woman. When the dominant follicles reached 18-20 mm, HCG 10000 was administered. Three D power Doppler US was done for every woman at the day after HCG administration. Ovum pick up was done after 35 hours following HCG administration. The luteal phase was supported by progesterone 300 mg per day . Five days following ovum pick up, the embryos were transferred at the blastocyst stage.
  Interventions: Diagnostic Test: 3D power doppler US

INTERVENTIONS:
Diagnostic Test: 3D power doppler US — Three D power Doppler US was done for every woman at the day after HCG administration. Ovum pick up was done after 35 hours following HCG administration.

SUMMARY:
Three D power Doppler US was done for every woman at the day after HCG administration. Ovum pick up was done after 35 hours following HCG administration. The luteal phase was supported by progesterone 300 mg per day (progest, micronized progesterone 100mg, Technopharma, Egypt, for pharco pharmaceuticals, Amriya- Alexandria). Five days following ovum pick up, the embryos were transferred at the blastocyst stage.

DETAILED DESCRIPTION:
All women underwent long agonist protocol for controlled ovarian hyperstimulation described by Chang et al. (14) The GnRH agonist was started in the previous mid-luteal phase (decapeptylR R 0.1mg, Triptorelin-Acetate, Ferring GmbH, Wittland 11, D-24109, and Kiel, Germany). After the confirmation of pituitary down regulation (serum LH less than 5 m IU/ml and serum E2 less than 50 pg /ml), the HMG ampoules were started by 225 IU/day (Gonapure 75 IU, IBSA Institute Biochimique SA, Switzerland). During the follow up of overstimulation, the doses were adjusted according to the response of patient. All women underwent serial TVS until at least three dominant follicles were reached in every woman. When the dominant follicles reached 18-20 mm, HCG 10000 (Choriomon 5000 IU, IBSA Institute Biochimique SA, Switzerland) was administered. Three D power Doppler US was done for every woman at the day after HCG administration. Ovum pick up was done after 35 hours following HCG administration. The luteal phase was supported by progesterone 300 mg per day (progest, micronized progesterone 100mg, Technopharma, Egypt, for pharco pharmaceuticals, Amriya- Alexandria). Five days following ovum pick up, the embryos were transferred at the blastocyst stage. Twelve days later to embryo transfer, serum pregnancy test was done and if positive (chemical pregnancy), the clinical pregnancy was confirmed by TVS for detection of gestational sacs and embryo cardiac activity. The ongoing pregnancy was detected by abdominal ultrasound at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

a

* age; 22-35 years,
* BMI; less than 35 kg/m2,
* Husband with oligo- or oligoasthenospermia.

Exclusion Criteria:

* \1-gross uterine and tubal pathology,
* 2-Development of OHSS,
* 3-poor responders,
* 4-failure of oocyte fertilization or failure of the embryos to reach the blastocyst stage and
* 5-Refusal to participate in the study at any step of the ICSI cycle.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: infertile women in need for ICSI due to male factor
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
chemical pregnancy | 14 day
  positive pregnancy test
the clinical pregnancy | 28 day
  was confirmed by TVS for detection of gestational sacs and embryo cardiac activity.
The ongoing pregnancy | 3 months
  was detected by abdominal ultrasound at 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: khalid salama, Principal Investigator — Benha University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ledee-Bataille N, Lapree-Delage G, Taupin JL, Dubanchet S, Frydman R, Chaouat G. Concentration of leukaemia inhibitory factor (LIF) in uterine flushing fluid is highly predictive of embryo implantation. Hum Reprod. 2002 Jan;17(1):213-8. doi: 10.1093/humrep/17.1.213. PMID 11756390